CLINICAL TRIAL: NCT03673800
Title: Cognitive Control Training in Online Problem Gambling: an Online Randomized Controlled Trial Among Non-treatment Seeking Problem Gamblers
Brief Title: Cognitive Control Training in Online Problem Gambling
Acronym: TRAIN-ONLINE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ARJEL (Autorité de Régulation des Jeux En Ligne) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P170601; 2017-A01666-47 (Other: IDRCB)
Record Dates: First submitted 2018-08-27; First posted 2018-09-17 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Pathological Gambling
Keywords: gambling disorder; pathological gambling; problem gambling; addiction
MeSH Terms: conditions — Gambling; Behavior, Addictive | interventions — Cognitive Training; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): Online Cognitive training on the Scientific Brain Training® (SBT®) platform with optional guidance by phone
  Interventions: Other: Experimental Group
- Online sensorial program (Sham Comparator): Online sensorial program on the Scientific Brain Training® (SBT®) platform with optional guidance by phone
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental Group — Cognitive web-based training : 2 up to 30 minutes sessions a week during 6 weeks. Optional debriefing by a neuropsychologist up to 15 minutes twice a week
  Other Names: Cognitive training with optional guidance by phone
  Arms: Cognitive Training
Other: Control Group — Sensorial web-based training : 2 up to 30 minutes sessions a week during 6 weeks. Optional debriefing by a neuropsychologist up to 15 minutes twice a week
  Arms: Online sensorial program

SUMMARY:
An online single blinding, randomized, comparative therapeutic web-based, controlled trial. The main objective of the study is to assess the clinical efficacy of an online computerized cognitive training program targeted on cognitive control, namely on inhibition, measured with the PGSI-recent, a modified version of Problem Gambling Severity Index (PGSI) with a 30 days recall period in patients with problem gambling, at 6 weeks, as compared to a control program with a similar setting.

DETAILED DESCRIPTION:
Cognitive training is currently used in brain damaged patients and in some psychiatric conditions, like schizophrenia or depression. Very few cognitive training programs have been published and tested in addictive disorders.

Training online is currently proposed in standard care, and is listed as recommended activities in daily hospitalization in addiction specialized out-settings in France.

The purpose of this research is to test the efficacy of an online intervention in gambling addiction through cognitive training targeting cognitive control inhibition.

The experimental Intervention (Cognitive Training) is a computerized cognitive training targeting inhibitory control of motor response (Scientific Brain Training®).The tasks included in the program have been selected and modified to target inhibition.

Control intervention is a sensorial program with a similar format targeting visual acuity. This is not a cognitive program, and can be considered as neutral in the addiction field.

An optional guidance by phone performed by a trained neuropsychologist is proposed to the included subjects in both groups, up to15 minutes twice a week.

Study design: A therapeutic web-based, comparative, randomized controlled trial, 2 arms, single blinding, with 52 weeks follow-up:

* a 14 weeks patient follow up (6 weeks for efficacy assessment and maintenance at 14 weeks).
* 52 weeks gambling account based data extracted from the ARJEL database in last 4 weeks before baseline, week 6, week 14 and week 52.

Population of study participants : Problem gamblers who will contact the responsible of the study.

Schedule for the study :

* Duration of inclusion period: 8 months
* Duration of patient participation: 52 weeks (12 months) including 14 weeks of active gambler participation and up to 52 weeks for the collection of gambler data from the ARJEL database.
* Total research duration: 20 months Main objective : To assess the clinical efficacy of an online computerized cognitive training program targeted on cognitive control, namely on inhibition, measured with the PGSI-recent, a modified version of Problem Gambling Severity Index (PGSI) with a 30 days recall period in patients with problem gambling, at 6 weeks.

Secondary objectives of the study are:

* to assess the efficacy on the evolution of the gambling behaviour assessed by the account player based gambling data, at 6, 14and 52 weeks.
* to assess the efficacy on the evolution of the self-reported gambling practice, and of quality of life at 0, 6 and 14 weeks.
* to assess the efficacy on the evolution of inhibition performance at the neuropsychological level at 0, 6 and 14, weeks.
* We will also assess the acceptability of this program and the preferred level of guidance of the non-treatment seeking problem gamblers as factor of response.

Statistical analysis:The change in PGSI-recent total score over 6 weeks will be compared with the student's t-test. If the test application conditions are not met, a Wilcoxon test will be applied.

ELIGIBILITY:
Inclusion criteria

1. Over 18 years old gamblers
2. Willing to share his/her first name, last name, exact birthdate, and exact place of birth (city + department). These informations are needed to extract ARJEL player account based gambling data, to avoid any doubloon or homonym.
3. PGSI-recent ≥ 5.
4. Recipient or beneficiary of the French social security system and resident in France.

Non-inclusion criteria

1. Gamblers cannot speak or understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The change over 6 weeks in Problem gambling severity index (PGSI)-recent total score, collected by internet | Change from baseline at 6 weeks
  PGSI-recent, a modified version of Problem Gambling Severity Index (PGSI) with a 30 days recall period in patients with problem gambling, at 6 weeks

SECONDARY OUTCOMES:
Problem gambling severity index - recent (PGSI) | Between baseline (T0) , and 14 weeks (T2)
Short form of Urgency, Premeditation, Perseverance, Sensation seeking, and Positive urgency (UPPS-P) Impulsive behavior scale | Between baseline (T0) , 6 weeks (T1) and 14 weeks (T2)
  Impulsivity scale
Time Line Follow Back (TLFB) -gambling | Between baseline (T0) , 6 weeks (T1) and 14 weeks (T2)
  Money and time spent gambling including offline gambling
EuroQol five dimensions questionnaire (EQ-5D) | Between baseline (T0) , 6 weeks (T1) and 14 weeks (T2)
  Health related quality of life self-questionnaire
Gambling Quality of Life Scale (GQoLS) | Between baseline (T0) , 6 weeks (T1) and 14 weeks (T2)
  Health related quality of life self-questionnaire specific to gambling disorder
Neuropsychological assessment: Stop Signal Task (SST) | Between baseline (T0) , 6 weeks (T1) and 14 weeks (T2)
  Cognitive task assessing inhibition
Total Deposit | In last 4 weeks before baseline (T0) , 6 weeks (T1), 14 weeks (T2) and 52 weeks (T3)
  Total Deposit assessed by the account player based gambling data (ARJEL database)
Total stake by game | In last 4 weeks before baseline (T0) , 6 weeks (T1), 14 weeks (T2) and 52 weeks (T3)
  Total stake by game assessed by the account player based gambling data (ARJEL database)
Compulsivity | In last 4 weeks before baseline (T0) , 6 weeks (T1), 14 weeks (T2) and 52 weeks (T3)
  Compulsivity (as defined by three consecutive deposits in a 12-hour period of time) assessed by the account player based gambling data (ARJEL database)
Number of deposit in the hour following a stake | In last 4 weeks before baseline (T0) , 6 weeks (T1), 14 weeks (T2) and 52 weeks (T3)
  Number of deposit in the hour following a stake assessed by the account player based gambling data (ARJEL database)
Total loss by game | In last 4 weeks before baseline (T0) , 6 weeks (T1), 14 weeks (T2) and 52 weeks (T3)
  Total loss by game assessed by the account player based gambling data (ARJEL database)
Number of sessions (all games) | In last 4 weeks before baseline (T0) , 6 weeks (T1), 14 weeks (T2) and 52 weeks (T3)
  Number of sessions (all games) in a clinical meaning assessed by the account player based gambling data (ARJEL database) Session is defined as gambling behaviour in itself; we'll consider the beginning of a session when a gambling action occurs after no gambling action since at least 30 minutes, and the end of the gambling session a gambling action followed by no gambling action during 30 minutes.
Session duration (poker only) | In last 4 weeks before baseline (T0) , 6 weeks (T1), 14 weeks (T2) and 52 weeks (T3)
  Session duration (poker only) assessed by the account player based gambling data (ARJEL database)
Gambling time slot | In last 4 weeks before baseline (T0) , 6 weeks (T1), 14 weeks (T2) and 52 weeks (T3)
  Gambling time slot assessed by the account player based gambling data (ARJEL database).
  The time slots are divided as follows:
  1. 0:00 to 3 :59
  2. 4:00 to 7:59
  3. 8:00 to 11:59
  4. 12:00 to 15:59
  5. 16:00 to 19:59
  6. 20:00 to 23:59
Acceptability of the online program assessed by the number of training session | At 6 week (T1)
Acceptability of the online program assessed by the length of training session | At 6 week (T1)
Level of guidance assessed by the number of phone session | At 6 week (T1)
  Number of debriefing by phone sessions
Level of guidance assessed by the length of phone session | At 6 week (T1)
  Length of debriefing by phone sessions

CONTACTS AND LOCATIONS:
Overall Officials: Amandine LUQUIENS, MD, PhD, HDR, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- Paul Brousse Hospital, Villejuif, France

REFERENCES:
- [Derived] Santiago A, Carre A, Miranda R, Lemogne C, LeStrat Y, Benyamina A, Perney P, Luquiens A. Study protocol for an online randomised controlled trial among non-treatment seeking problem gamblers: training inhibition in online problem gambling (TRAIN-online) trial. BMJ Open. 2021 Nov 30;11(11):e051641. doi: 10.1136/bmjopen-2021-051641. PMID 34848517